CLINICAL TRIAL: NCT05214534
Title: Contribution of SuPAR for Patients in a Situation of Uncertainty Downstream of Emergencies
Acronym: SuPAR
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 MOUSTAFA; 2021-A01930-41 (Other: 2021-A01930-41)
Record Dates: First submitted 2021-12-08; First posted 2022-01-28 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2021-11

CONDITIONS: Emergencies; Disease; In-hospital Observation
Keywords: Supar; Patient triage; Emergency
MeSH Terms: conditions — Emergencies; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — bottoms of the of blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Retrospective analysis of the correlation between SuPAR measurement and patient outcome after hospitalization
  Interventions: Other: blood supar measurement

INTERVENTIONS:
Other: blood supar measurement — The supar values will be measured afterwards on the tube bottoms of the patients included in the study from their usual collection

SUMMARY:
In this study, the investigators will investigate the relationship between the blood level of SuPAR at admission to the emergency department of the Clermont-Ferrand University Hospital, and the outcome of patients after their hospitalization in a short stay unit.

DETAILED DESCRIPTION:
SuPAR (Soluble urokinase Plasminogen Activator Receptor) is a non-specific prognostic blood biomarker related to inflammation. An elevated SuPAR value reflects significant chronic inflammation and predicts a risk of negative outcome and even short-term mortality (intra-hospital, 30 days, 90 days). Conversely, a low SuPAR value is a strong indicator of good prognosis and low risk of readmission. It is therefore of interest to know a patient's SuPAR blood level to enable the clinician to decide whether the patient should be admitted or discharged. SuPAR has been shown to be the best prognostic marker associated with the presence and progression of disease and risk of mortality. The use of SuPAR in clinical routine adds significant complementary information to the standard Early Warning Score assessment and to the classical parameters such as CRP, PCT, Lactate, ALT, Bilirubin, and CBC in the pre-admission of acute patients.

Patients admitted to the emergency department will receive their usual management. We will test the added value of the SuPAR assay in the prognosis of patients' outcome at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years old
* Admitted to the emergency department of the Clermont-Ferrand University Hospital for a medical reason,
* Classified as FRENCH II or III by the nurse organizer of the reception management
* Necessity of clinical observation in the Short Term Hospitalization Unit for final orientation decision
* Requires a blood test upon arrival in the emergency department
* Able to give informed non-opposition to participate in the research.
* Affiliation to a Social Security system

Exclusion Criteria:

* Patient under guardianship or curatorship
* Pregnant and breast feeding woman
* Patient admitted for psychiatric pathology
* Patient with a limitation of therapeutics
* Refusal to participate
* Patient hospitalized because of a particular social context

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients requiring clinical observation for a final referral decision and meeting the eligibility criteria will be offered the study
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Relationship between blood supar levels and patient outcome at discharge | When the excepted 150 patients will be included, estimated 6 months
  Relation between blood supar levels measured and patient outcome at discharge evaluated as : return home = good evolution; hospitalization = bad evolution; admission to an intensive care unit or death = unfavorable evolution

SECONDARY OUTCOMES:
National Early Warning Score 2 (NEWS2) | Hour 0
  Score allowing the classification of the urgency of a patient. The minimum value is 0 and the maximum value is 20. Higher scores mean a worse outcome
Modified Early Warning Score (MEWS) | Hour 0
  Score allowing the classification of the urgency of a patient. The minimum value is 0 and the maximum value is 17. Higher scores mean a worse outcome
Blood supar levels | When the excepted 150 patients will be included, estimated 6 months
  the supar values are classifies into three categories : < 3 ng/ml : supports the referral decision. the patient's general condition is good and the prognosis is high 3-6 ng/ml : presence of pathologies and comorbidity factors. readmissions and high mortality beyond 6 months >6 ng/ml : requires special clinical attention, high risk of mortality
Blood CRP value | Hour 0
  the CRP value will be assessed during the blood test performed as part of the classical management when the patient arrives in the emergency room
Cardiac frequency | Hour 0
  cardiac frequency will be evaluated when the patient arrives in the emergency service as part of the classical management
Respiratory rate | Hour 0
  respiratory rate will be evaluated when the patient arrives in the emergency service as part of the classical management
Temperature | Hour 0
  the temperature will be evaluated when the patient arrives in the emergency service as part of the classical management
Systolic blood pressure | Hour 0
  systolic blood pressure will be evaluated when the patient arrives in the emergency service as part of the classical management
Diastolic blood pressure | Hour 0
  diastolic blood pressure will be evaluated when the patient arrives in the emergency service as part of the classical management
French triage | Hour 0
  French Emergency Nurses Classification in Hospitals (FRENCH) ranks priorities from 5 to 1 (from least urgent to most urgent) according to prognosis and complexity/severity of the medical condition
Main diagnosis retained by the physician | at the end of hospitalization
  Main diagnosis retained

CONTACTS AND LOCATIONS:
Overall Officials: Farès Moustafa, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France